CLINICAL TRIAL: NCT01949285
Title: A Theranostic Tool to Assess and Enable Spared Spinal Motor Function After SCI
Brief Title: Transcutaneous Electrical Spinal Cord Stimulation for Lower Limbs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroEnabling Technologies, Inc. (Industry)
Collaborators: University of California, Los Angeles (Other); California Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NETI201309
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-04

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; Paralysis; Rehabilitation; Assessment; Theranostics
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grp#1: sham stimulation (Sham Comparator): Group #1: Baseline clinical assessment; followed by two weeks training with no stimulation; then four weeks training + sham Transcutaneous Electrical Spinal Cord Stimulation; followed by repeat clinical assessment; then four weeks training + effective non-sham Transcutaneous Spinal Cord Stimulation; repeat clinical assessment.
  Secondary outcome measurements: assess ability to stand with and without stimulation using a stance frame support; assess trunk function (core stability) with and without stimulation
  Interventions: Device: Transcutaneous Electrical Spinal Cord Stimulation
- Grp#2: Control (Active Comparator): Group #2: Baseline clinical assessment; followed by two weeks training with no Transcutaneous Electrical Spinal Cord Stimulation; then four weeks training + effective Transcutaneous Electrical Spinal Cord Stimulation; followed by repeat clinical assessment.
  Secondary outcome measurements: assess ability to stand with and without stimulation using a stance frame support; assess trunk function (core stability) with and without stimulation
  Interventions: Device: Transcutaneous Electrical Spinal Cord Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Spinal Cord Stimulation — A prototype device that non-invasively delivers electrical stimulation to the spinal cord will be used to assess and rehabilitate spared spinal cord function.
  Other Names: Prototype Device

SUMMARY:
This study is to determine if non-invasive electrical stimulation of the spinal cord can be used to: 1) assess spared function following a spinal cord injury; and 2) be use for rehabilitation.

DETAILED DESCRIPTION:
This study is to determine if non-invasive electrical stimulation of the spinal cord can be used to: 1) assess spared function following a spinal cord injury; and 2) be use for rehabilitation.

The investigators hypothesize that this type of stimulation can be used to locate and determine if any spinal (nerve) pathways or connections were spared following a spinal cord injury. We also hypothesize the same stimulation can help revive or recover function to muscles connected to these spared spinal (nerve) pathways in individuals who are clinically paralyzed. Our research has demonstrated that modifying the activation state of the spinal cord after an injury, or awakening the spinal cord, can benefit people with paralysis years after a spinal cord injury. This method and device have not yet been approved by the FDA for the treatment of paralysis and are under investigation. This study if successful will help provide further evidence that could be use to one day to gain FDA approval.

ELIGIBILITY:
Inclusion Criteria: SCI ASIA A, B, C

* Spinal cord injury 1 or more years prior
* Non progressive cervical or thoracic SCI
* Half of key muscles below neurological level having a motor score of less than 2/5
* Ability to commit to home exercises and 16 week participation
* Stable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate participation in lower extremity rehabilitation or testing activities
* Not dependent on ventilation support
* No painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or urinary tract infection that might interfere with lower extremity rehabilitation or testing activities
* No clinically significant depression or ongoing drug abuse
* Adequate social support network to be able to participate in weekly training and assessment sessions for the duration of the 16 week study period
* No current anti-spasticity regimen
* Must not have received botox injections in the prior six months
* Be unable to use lower extremity for functional tasks

Exclusion Criteria:

* Pregnancy
* No functional segmental reflexes below the lesion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in sensorimotor function in the lower extremities | 10-12 weeks
  Subjects will be tested by several measures of sensory and motor function, as well as self assessments of spasticity, quality of life, and independence. These tests include:
  American Spinal Injury Association (ASIA) scoring system, Spinal Cord Independence Measure (SCIM), Ashworth Spasticity Scale, Penn Spasm Frequency, Visual Analog Scale (VAS) for Spasticity, Electromyographic (EMG) recordings, Joint angle (goniometer) measures, kinematic analysis.

SECONDARY OUTCOMES:
Ability to stand independently | 2-4 weeks
  Subjects will be evaluated on their core body function and ability to stand

CONTACTS AND LOCATIONS:
Overall Officials: Victor R Edgerton, PhD, Study Chair — University of California, Los Angeles; Nicholas A Terrafranca, DPM, Principal Investigator — NeuroEnabling Technologies, Inc.
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States